CLINICAL TRIAL: NCT03154242
Title: Effect of Genetic Polymorphisms on Clinical Outcome of Platinum Based Chemotherapy in Non-Small Cell Lung Cancer Patients
Brief Title: Effect of Genetic Polymorphisms on Platinum Based Chemotherapy in Non Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Esraa Salah Abdal Hay Abdal Khalek, demonstrator of clinical pharmacy, Ain Shams University
Other Study IDs: PHCL137
Record Dates: First submitted 2017-05-09; First posted 2017-05-16 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: non small cell lung cancer; NSCLC; Platinum
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Device: No | US Export: No

SUMMARY:
This Study evaluate the effect of Polymorphism in the Excision repair cross-complementing group 5 (ERCC5) (rs1047768 and rs751402) gene on the clinical outcome of Platinum-based regimens used in the treatment of Non-Small Cell Lung Cancer (NSCLC) patients

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with immunohistochemically and pathologically confirmed non-small cell lung cancer (NSCLC).
2. Eastern Cooperative Oncology Group performance status (ECOG PS) = 0-2.
3. Chemotherapy naïve.
4. Age >18 years.
5. Adequate bone marrow reserve

Exclusion Criteria:

1. Presence of Central nervous system(CNS) metastases.
2. Inadequate liver function
3. Inadequate renal function
4. Serious comorbid systemic disorder incompatible with the study.
5. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical oncology department at Al Demerdash hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the date of starting the chemotherapy until the date of documented disease progression or date of death from any cause assessed up to 12 months
  It's defined as the time from day 1 of chemotherapy to the day of documented disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Esraa S Abdalkhalek, Principal Investigator — Ain Shams University
Locations (1):
- Al Demerdash Hospital, Cairo, Egypt